CLINICAL TRIAL: NCT02437006
Title: Early Intervention With a Low-intensity Leg Cycling Exercise Program for Individuals After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: KMUH-IRB- 20130376
Record Dates: First submitted 2015-03-31; First posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2014-03

CONDITIONS: Stroke
Keywords: stroke; exercise capacity
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rehabilitation (No Intervention): half an hour physical and half an hour occupational therapy in rehabilitation
- Low-intensity exercise (Experimental): Low-intensity exercise plus rehabilitation
  Interventions: Other: exercise
- High-intensity exercise (Experimental): High-intensity exercise plus rehabilitation
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — cycle ergometry
  Arms: High-intensity exercise; Low-intensity exercise

SUMMARY:
This is a two-stage study. In the first stage, 30 subjects with stroke (onset > 2 weeks) are recruited, and they are assessed and recorded with clinical characteristics, sympathetic nerve testing, and twice symptom-limit exercise capacity tests. The second stage would recruited 90 subjects with stroke (onset>2 weeks), and they are randomized to one of three groups (control, low-intensity, high-intensity). They are evaluated before and after the four-week interval with clinical characteristics and twice symptom-limit exercise capacity tests (baseline and after four-week training) .

DETAILED DESCRIPTION:
This is a two-stage study. In the first stage, 30 subjects with stroke (onset > 2 weeks) are recruited, and they are assessed and recorded with sympathetic nerve testing, anthropometry, and twice symptom-limit exercise capacity tests.The second stage would recruited 90 subjects with stroke (onset>2 weeks), and they are randomized to one of three groups. The control group undergoes traditional rehabilitation only, The low-intensity exercise group receives a low-intensity four-week cycle ergometry and traditional rehabilitation. The The high-intensity exercise group gets a high-intensity four-week cycle ergometry and traditional rehabilitation. They are evaluated by sympathetic tests, anthropometry, functional scales and activity questionnaires, and symptom-limit exercise capacity tests before and after the four-week training.

ELIGIBILITY:
Inclusion Criteria:

* stroke onset longer than two weeks,
* eligible for exercise testing by Doctor

Exclusion Criteria:

* aphasia,
* apraxia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
change values of symptom-limit exercise capacity | baseline and after four-week training
  value was showed by oxygen uptake (mL/kg/min)

SECONDARY OUTCOMES:
change values of sympathetic nerve tests | baseline and after four-week training
  change value was measure by blood pressure (from lying to stand, mm-Hg) at baseline and after four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miao-Ju Hsu, PHD, Principal Investigator — Kaohsiung Medical University, College of Health Sciences
Locations (1):
- Kaohsiung Medical University, College of Health Sciences, Kaohsiung City, Taiwan